CLINICAL TRIAL: NCT06222008
Title: Correlation Study of Symptom Clusters and Negative Emotions During Chemotherapy in Ovarian Cancer Patients With Different Chinese Medicine Constitution
Brief Title: Study on Symptom Clusters During Chemotherapy in Ovarian Cancer Patients With Different Chinese Medicine Constitution
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yandi Zhu (Other)
Responsible Party: Sponsor-Investigator, Yandi Zhu, Associate Chief Nurse, Affiliated Hospital of Jiaxing University
Organization: Affiliated Hospital of Jiaxing University (Other)
Other Study IDs: FirstHJiaxing01
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Radiotherapy Side Effect; Symptom Cluster
MeSH Terms: conditions — Ovarian Neoplasms; Radiation Injuries; Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no Intervention — Observational study, no intervention

SUMMARY:
The goal of this observational study is to learn about in Patients treated with postoperative chemotherapy for ovarian tumors. The main questions it aims to answer are: • [What symptom clusters are present in patients treated with postoperative chemotherapy for ovarian tumors] • [Are there differences in symptom clusters for patients with different TCM body types] Participants will [complete questionnaires prior to the start of chemotherapy and after the 1st, 3rd, and 6th chemotherapy treatments].

ELIGIBILITY:
Inclusion Criteria:

Pathologic diagnosis of ovarian cancer, the treatment plan adopts surgery combined with chemotherapy.

Age ≥ 18 years old, know the real situation of the disease, the expected survival period > 1 year.

General condition is good, no history of psychiatric disease, no serious heart, brain, liver, kidney function abnormality.

Informed consent and voluntarily participate in this study.

Exclusion Criteria:

those who have other tumors or whose diagnosis is unclear. those who cannot communicate properly, understand the questionnaire or complete the scale assessment.

those who receive additional psychological interventions during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients with ovarian malignant tumors undergoing chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy Symptoms | Average 1 year
  Symptoms during chemotherapy,Examples include nausea, vomiting, hair loss, fatigue , etc.

SECONDARY OUTCOMES:
Chemotherapy symptom clusters | Average 1 year
  The internal consistency, content validity, and validity of the scale were verified by combining the 13 core symptom items in the Chinese Version of the M.D. Anderson Symptom Inventory (MDASI-C) with the 9 ovarian cancer-specific symptoms. All entries (22) are numbered "0" to "10" to represent the degree of symptoms from "nonexistent" to "worst imaginable", and the symptoms assessed ranged from "nonexistent" to "worst imaginable". "The onset of the assessed symptoms was limited to the last 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jiaxing, Jiaxing, China

IPD SHARING:
Plan to Share IPD: No